CLINICAL TRIAL: NCT05940961
Title: A Multicenter Prospective Clinical Study of Inotuzumab Ozogamicin (INO) in the Treatment of Minimal Residual Disease Recurrent After Hematopoietic Stem Cell Transplantation of Acute Lymphoblastic Leukemia (ALL)
Brief Title: Inotuzumab Ozogamicin in the Treatment of MRD+ After HSCT of ALL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sheng-Li Xue, MD (Other)
Collaborators: Jining Medical University (Other); The Second People's Hospital of Huai'an (Other); The First Affiliated Hospital of Bengbu Medical University (Other); Affiliated Hospital of Nantong University (Other); Suzhou Hospital of Traditional Chinese Medicine (Other); Northern Jiangsu People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Sheng-Li Xue, MD, Professor, The First Affiliated Hospital of Soochow University
Organization: The First Affiliated Hospital of Soochow University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: szINO
Record Dates: First submitted 2023-07-01; First posted 2023-07-11 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: ALL; MRD-positive; Hematopoietic Stem Cell Transplantation
MeSH Terms: interventions — Inotuzumab Ozogamicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inotuzumab Ozogamicin in the Treatment of MRD+ After HSCT of ALL (Experimental): intravenous infusion: Cycle 1: D1 0.8mg/m2, D8 0.5mg/m2, D15 0.5mg/m2, if the MRD turn negative, cycle 2: D1 0.5mg/m2, D8 0.5mg/m2, D15 0.5mg/m2， if not，cycle 2: D1 0.8mg/m2, D8 0.5mg/m2, D15 0.5mg/m2
  Interventions: Drug: Inotuzumab Ozogamicin

INTERVENTIONS:
Drug: Inotuzumab Ozogamicin — intravenous infusion: Cycle 1: D1 0.8mg/m2, D8 0.5mg/m2, D15 0.5mg/m2, if the MRD turn negative, cycle 2: D1 0.5mg/m2, D8 0.5mg/m2, D15 0.5mg/m2， if not，cycle 2: D1 0.8mg/m2, D8 0.5mg/m2, D15 0.5mg/m2
  Other Names: INO

SUMMARY:
As part of postremission consolidative therapy, the decision to proceed with hematopoietic stem cell transplantation is a recommendable regimen in ALL therapy. However, The recurrence rate is high after transplantation. Minimal Residual Disease (MRD) is an important factor affecting the effect of HSCT. The hematologic recurrence rate of MRD-positive patients with adult ALL is high.

MRD- is associated with better prognosis. Therefore, maintaining MRD- after transplantation is necessary for long-term survival. The purpose of this study is to explore the efficacy and safety of Inotuzumab Ozogamicin in the treatment of minimal residual disease recurrence after HSCT of ALL patients.

DETAILED DESCRIPTION:
As part of postremission consolidative therapy, the decision to proceed with hematopoietic stem cell transplantation is a recommendable regimen in ALL therapy. However, The recurrence rate is high after transplantation. Minimal Residual Disease (MRD) is an important factor affecting the effect of HSCT. The hematologic recurrence rate of MRD-positive patients with adult ALL is high.

MRD- is associated with better prognosis. Therefore, maintaining MRD- after transplantation is necessary for long-term survival. INO-VATE confirmed that Inotuzumab Ozogamicin can be used to achieve high remission (CR/CRi) and MRD-negative rates, serving as an effective bridge to HSCT, and it is associated with increased OS and PFS in patients with R/R BCP ALL. The purpose of this study is to explore the efficacy and safety of Inotuzumab Ozogamicin in the treatment of minimal residual disease recurrence after HSCT of ALL patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 15 and ≤ 65 years.
2. Patients diagnosed with CD22+ B-ALL according to 2023 NCCN Acute Lymphoblasts Leukaemias diagnosis standard.
3. CD22+ B-ALL patients with MRD recurrence after HSCT. Ph+ ALL patients were eligible if treatment with 1 or more second-generation BCR::ABL1 tyrosine kinase inhibitors (TKIs) had failed,
4. ECOG performance status score less than 3.
5. Expected survival time #3 months.
6. Patients without serious heart, lung, liver, or kidney disease.
7. Ability to understand and voluntarily provide informed consent.

Exclusion Criteria:

1. Patients who are allergic to the study drug or drugs with similar chemical structures.
2. Pregnant or lactating women, and women of childbearing age who do not want to practice effective methods of contraception.
3. Active infection.
4. Active bleeding.
5. Patients with new thrombosis, embolism, cerebral hemorrhage, or other diseases or a medical history within one year before enrollment.
6. Patients with mental disorders or other conditions whereby informed consent cannot be obtained and where the requirements of the study treatment and procedures cannot be met.
7. Liver function abnormalities (total bilirubin > 1.5 times the upper limit of the normal range, ALT/AST > 2.5 times the upper limit of the normal range or patients with liver involvement whose ALT/AST > 1.5 times the upper limit of the normal range), or renal anomalies (serum creatinine > 1.5 times the upper limit of the normal value).
8. Patients with a history of clinically significant QTc interval prolongation (male > 450 ms; female > 470 ms), ventricular heart tachycardia and atrial fibrillation, II-degree heart block, myocardial infarction attack within one year before enrollment, and congestive heart failure, and patients with coronary heart disease who have clinical symptoms and requiring drug treatment.
9. Surgery on the main organs within the past six weeks.
10. Drug abuse or long-term alcohol abuse that would affect the evaluation results.
11. Patients who have received organ transplants (excepting bone marrow transplantation).
12. Patients not suitable for the study according to the investigator's assessment.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
the rate of MRD- | At the end of Cycle 1 and Cycle 2(each cycle is 21 days)
  For Ph-negative ALL: undetectable MRD by flow cytometry At the end of Cycle 1 and Cycle 2 (each cycle is 21 days) . For Ph-positive ALL: undetectable MRD by flow cytometry and absence of quantifiable BCR::ABL1 transcript by PCR At the end of Cycle 1 and Cycle 2(each cycle is 21 days).

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 1 year
  It is measured from the date of entry into this trial to the date of progression or death
Overall survival (OS) | 1 year
  It is measured from the date of entry into this trial to the date of death from any cause; patients not known to have died at last follow-up are censored on the date they were last known to be alive.
Adverse events in hematological system | 1 year
  Record of adverse events in hematological system during and after designed venetoclax combined azacitidine regimen induction
Adverse events in other organs or systems | 1 year
  Record of adverse events in other organs or systems during and after designed venetoclax combined azacitidine regimen induction.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No